CLINICAL TRIAL: NCT04890847
Title: A Platform for Multidisciplinary Medical Artificial Intelligence Development
Acronym: AI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Sun Yat-sen University
Other Study IDs: AIplatform-2020
Record Dates: First submitted 2021-03-18; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Medical Artificial Intelligence; Medical Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- human-machine collaboration group: healthcare professionals and machine collaboration for annotation and AI model development
- pure mannual group: healthcare professionals for pure manual annotation and AI model development

SUMMARY:
Biomedical deep learning (DL) often relies heavily on generating reliable labels for large-scale data and highly technical requirements for model training. To efficiently develop DL models, we established an integrated platform to introduce automation to both annotation and model training-the primary process of DL model development. Based on this platform, we quantitively validated and compared the annotation strategy and AI model development with the pure manual annotation method performed on medical image datasets from multiple disciplines.

ELIGIBILITY:
Inclusion Criteria:

* have medical imaging record (including ophthalmology, pathology, radiography, blood cells, and endoscopy)

Exclusion Criteria:

* unqualified medical imaging

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: medical imaging for multiple disciplines including ophthalmology, pathology, radiography, blood cells, and endoscopy
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
annotation accuracy | baseline
  calculate annotation accuracy for comparison between groups with using the annotation results

SECONDARY OUTCOMES:
accuracy of model performance | baseline
  calculate AI model accuracy for comparison between groups with using the model predicted results
AUC of model performance | baseline
  calculate AI model AUCs for comparison between groups with using the model predicted results
annotation time cost | baseline
  calculate annotation time cost for comparison between groups with using the time recorded during the tests

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, Ph.D, M.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen Univerisity
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen Univerisity, Guangzhou, Guangdong, China